CLINICAL TRIAL: NCT00881712
Title: A Phase II Trial of 3 Dimensional Proton Radiotherapy With Concomitant Chemotherapy for Patients With Initially Unresectable Stage III Non-Small Cell Lung Cancer
Brief Title: Proton Therapy With Chemotherapy for Stage III Non-Small Cell Lung Cancer (LU02)
Acronym: LU02
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: projected enrollment rate not feasible
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 0802-LU02
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Results first posted 2015-06-16 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-small cell lung Cancer; Proton Radiation; Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PET positive nodal disease measuring 15 mm or greater (Experimental): Proton radiation with concomitant chemotherapy
  Interventions: Radiation: PET positive nodal disease measuring 15 mm or greater
- PET positive nodal disease measuring less than 15 mm (Experimental): Proton radiation
  Interventions: Radiation: PET positive nodal disease measuring less than 15 mm
- Patients considered resectable (Experimental): Proton radiation plus surgery
  Interventions: Radiation: Patients considered resectable

INTERVENTIONS:
Radiation: PET positive nodal disease measuring 15 mm or greater — Proton radiation at 2 cobalt gray equivalent per fraction to a total of 74 cobalt gray equivalent with concomitant weekly chemotherapy.
  Other Names: Proton Radiation
  Arms: PET positive nodal disease measuring 15 mm or greater
Radiation: PET positive nodal disease measuring less than 15 mm — Proton radiation at 2 cobalt gray equivalent per fraction to a total of 60 cobalt gray equivalent with concomitant weekly chemotherapy.
  Other Names: Proton Radiation
  Arms: PET positive nodal disease measuring less than 15 mm
Radiation: Patients considered resectable — Proton radiation at 2 cobalt gray per fraction. Re-evaluation performed between days 18-22 of treatment. If considered resectable after re-evaluation, radiotherapy will discontinue after a total of 50 cobalt gray equivalent and surgery will be performed.
  Other Names: Proton Radiation
  Arms: Patients considered resectable

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, proton radiation at a higher tumor dose (and lower normal surrounding lung dose) combined with standard chemotherapy has on lung cancer. The dose you receive to the tumor will be higher than the standard dose. This may be able to increase the control of the tumor. Due to the accuracy of radiation given with protons, the dose to the normal lung tissue that surrounds the tumor will be lower than standard. This may be able to reduce the frequency and severity of the usual radiation side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented non-small cell carcinoma of the lung diagnosed within 16 weeks prior to study enrollment.
* Patient must be at least 18 years old at the time of consent.
* Stage III A or III B disease.
* Patients must be able to start study treatment within 6 weeks of study enrollment.
* Induction chemotherapy is allowed.
* Marginally resectable or unresectable at presentation.
* If the patient had exploratory thoracotomy, it must be done at least 3 weeks prior to enrollment.

Exclusion Criteria:

* Evidence of distant metastasis.
* Prior thoracic radiotherapy.
* Any history of allergic reaction to taxanes.
* Prior tumor resection. Candidate for upfront curative surgery.
* Pleural effusion visible on chest x-ray or the scout view of the CT chest.
* Unintentional weight loss within the month prior to diagnosis ≥ 10%.
* Previous or concomitant malignancy other than early stage tumor treated more than 3 years ago for cure.
* The presence of PET positive contralateral hilar disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradford S Hoppe, MD, MPH, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

REFERENCES:
- [Background] Cancer Facts and Figures 2008 - American Cancer Society http://www.cancer.org/downloads/STT/2008CAFFfinalsecured.pdf
- [Background] Delaney, Kooy editors: Proton and Charged particle Radiotherapy; LWW, 2008
- [Background] Chang JY, Zhang X, Wang X, Kang Y, Riley B, Bilton S, Mohan R, Komaki R, Cox JD. Significant reduction of normal tissue dose by proton radiotherapy compared with three-dimensional conformal or intensity-modulated radiation therapy in Stage I or Stage III non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):1087-96. doi: 10.1016/j.ijrobp.2006.01.052. Epub 2006 May 6. PMID 16682145
- [Background] Auberger T, Seydl K, Futschek T, Sztankay A, Sweeney RA, Lukas P. Photons or protons: precision radiotherapy of lung cancer. Strahlenther Onkol. 2007 Dec;183 Spec No 2:3-6. doi: 10.1007/s00066-007-2002-9. No abstract available. PMID 18166995
- [Background] Nichols RC, Henderson RH, Huh SN, Flampouri S, Cury JD, Pham DC, D'Agostino HJ, Louis D, Li Z, Mendenhall NP. Proton Radiotherapy Offers Reduced Bone Marrow and Normal Lung Exposure for Patients Receiving Dose Escalated Radiotherapy with Concomitant Chemotherapy for Regionally Advanced Non-Small Cell Lung Cancer. Presented at the LALCa 2008 - 3rd Latin American Conference on Lung Cancer - Tercera Conferencia Latinoamericana sobre Cancer Pulmonar - Vina del Mar, Chile - October 9 and 10, 2008
- [Background] Graham MV, Purdy JA, Emami B, Harms W, Bosch W, Lockett MA, Perez CA. Clinical dose-volume histogram analysis for pneumonitis after 3D treatment for non-small cell lung cancer (NSCLC). Int J Radiat Oncol Biol Phys. 1999 Sep 1;45(2):323-9. doi: 10.1016/s0360-3016(99)00183-2. PMID 10487552
- [Background] Lee HK, Vaporciyan AA, Cox JD, Tucker SL, Putnam JB Jr, Ajani JA, Liao Z, Swisher SG, Roth JA, Smythe WR, Walsh GL, Mohan R, Liu HH, Mooring D, Komaki R. Postoperative pulmonary complications after preoperative chemoradiation for esophageal carcinoma: correlation with pulmonary dose-volume histogram parameters. Int J Radiat Oncol Biol Phys. 2003 Dec 1;57(5):1317-22. doi: 10.1016/s0360-3016(03)01373-7. PMID 14630268
- [Background] Komaki R, Sejpal S, Wei X, et al. Reduction of Bone Marrow Suppression for Patients with Stage III NSCLC Treated by Proton and Chemotherapy Compared with IMRT and Chemotherapy. Proceedings of the PTCOG 47, May 19-24, 2008.
- [Background] Curran W, Scott C, Langer C, et al. Long term benefit is observed in a phase III comparison of sequential vs. concurrent chemo-radiation for patients with unresectable NSCLC: RTOG 9410. Proc Am Soc Clin Oncol 2003;61(abstr).
- [Background] Furuse K, Fukuoka M, Kawahara M, Nishikawa H, Takada Y, Kudoh S, Katagami N, Ariyoshi Y. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with mitomycin, vindesine, and cisplatin in unresectable stage III non-small-cell lung cancer. J Clin Oncol. 1999 Sep;17(9):2692-9. doi: 10.1200/JCO.1999.17.9.2692. PMID 10561343
- [Background] Rosenzweig KE, Sim SE, Mychalczak B, Braban LE, Schindelheim R, Leibel SA. Elective nodal irradiation in the treatment of non-small-cell lung cancer with three-dimensional conformal radiation therapy. Int J Radiat Oncol Biol Phys. 2001 Jul 1;50(3):681-5. doi: 10.1016/s0360-3016(01)01482-1. PMID 11395236
- [Background] Martel MK, et al. Incidental doses to clinically negative nodes from conformal treatment fields for non-small cell lung cancer. Int J Rad Oncol Biol Phys. 45(3 (supplement)): 244, 1999.
- [Background] Nichols RC, Huh SN, Hoppe BS, Henderson RH, Li Z, Mendenhall NP. Protons Safely Allow Coverage of High Risk Nodes for Patients with Regionally Advanced NSCLC, University of Florida Proton Therapy Institute. Submitted for consideration. American Radium Society, 2009.
- [Background] Rosenman JG, Halle JS, Socinski MA, Deschesne K, Moore DT, Johnson H, Fraser R, Morris DE. High-dose conformal radiotherapy for treatment of stage IIIA/IIIB non-small-cell lung cancer: technical issues and results of a phase I/II trial. Int J Radiat Oncol Biol Phys. 2002 Oct 1;54(2):348-56. doi: 10.1016/s0360-3016(02)02958-9. PMID 12243807
- [Background] Perez CA, Pajak TF, Rubin P, Simpson JR, Mohiuddin M, Brady LW, Perez-Tamayo R, Rotman M. Long-term observations of the patterns of failure in patients with unresectable non-oat cell carcinoma of the lung treated with definitive radiotherapy. Report by the Radiation Therapy Oncology Group. Cancer. 1987 Jun 1;59(11):1874-81. doi: 10.1002/1097-0142(19870601)59:113.0.co;2-z. PMID 3032394
- [Background] Fletcher GH. Clinical dose-response curves of human malignant epithelial tumours. Br J Radiol. 1973 Jan;46(541):1-12. doi: 10.1259/0007-1285-46-541-1. No abstract available. PMID 4630323
- [Background] Albain KS, Swann RS, Rusch VR, et al. Phase III study of concurrent chemotherapy and radiotherapy (CT/RT) vs. CT/RT followed by surgical resection for stage IIIA (pN2) non-small cell lung cancer (NSCLC): Outcomes update of North American Intergroup 0139 (RTOG 9309). Proc Am Soc Clin Oncol, abstract 7014, 2005.
- [Background] Lau D, Leigh B, Gandara D, Edelman M, Morgan R, Israel V, Lara P, Wilder R, Ryu J, Doroshow J. Twice-weekly paclitaxel and weekly carboplatin with concurrent thoracic radiation followed by carboplatin/paclitaxel consolidation for stage III non-small-cell lung cancer: a California Cancer Consortium phase II trial. J Clin Oncol. 2001 Jan 15;19(2):442-7. doi: 10.1200/JCO.2001.19.2.442. PMID 11208837
- [Background] Choy H, Akerley W, Safran H, Graziano S, Chung C, Williams T, Cole B, Kennedy T. Multiinstitutional phase II trial of paclitaxel, carboplatin, and concurrent radiation therapy for locally advanced non-small-cell lung cancer. J Clin Oncol. 1998 Oct;16(10):3316-22. doi: 10.1200/JCO.1998.16.10.3316. PMID 9779707
- [Background] Vokes E, Herndon J, Turrisi A. Induction chemotherapy followed by concomitant chemoradiotherapy (CT/XRT) versus CT/XRT alone for regionally advanced unresectable non-small cell lung cancer (NSCLC): Initial analysis of a randomized phase III trial. Pro Amer Soc Clin Oncol. 23(616A), 2004.
- [Background] Bradley J, et al. Phase I results of RTOG 0117; A phase I/II dose intensification study using 3DCRTand concurrent chemotherapy for patients with inoperable non-small cell lung cancer. Pro Amer Soc Clin Oncol. 24: p. 7063A, 2005.
- [Background] Blackstock A. Cancer and Leukemia Group B: Induction plus concurrent chemotherapy with high dose (74 Gy) 3 dimensional (3-D) thoracic radiotherapy in stage III non-small cell lung cancer. Preliminary report of CALGB 30105. Pro Amer Soc Clin Oncol. 24(1): 7042, 2006.
- [Background] Roth JA, Atkinson EN, Fossella F, Komaki R, Bernadette Ryan M, Putnam JB Jr, Lee JS, Dhingra H, De Caro L, Chasen M, Hong WK. Long-term follow-up of patients enrolled in a randomized trial comparing perioperative chemotherapy and surgery with surgery alone in resectable stage IIIA non-small-cell lung cancer. Lung Cancer. 1998 Jul;21(1):1-6. doi: 10.1016/s0169-5002(98)00046-4. PMID 9792048
- [Background] Belani CP, Choy H, Bonomi P, Scott C, Travis P, Haluschak J, Curran WJ Jr. Combined chemoradiotherapy regimens of paclitaxel and carboplatin for locally advanced non-small-cell lung cancer: a randomized phase II locally advanced multi-modality protocol. J Clin Oncol. 2005 Sep 1;23(25):5883-91. doi: 10.1200/JCO.2005.55.405. Epub 2005 Aug 8. PMID 16087941
- [Background] Chvetsov AV, Palta JJ, Nagata Y. Time-dependent cell disintegration kinetics in lung tumors after irradiation. Phys Med Biol. 2008 May 7;53(9):2413-23. doi: 10.1088/0031-9155/53/9/013. Epub 2008 Apr 17. PMID 18421118
- [Background] Chapet O, Kong FM, Quint LE, Chang AC, Ten Haken RK, Eisbruch A, Hayman JA. CT-based definition of thoracic lymph node stations: an atlas from the University of Michigan. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):170-8. doi: 10.1016/j.ijrobp.2004.12.060. PMID 16111586

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PET Positive Nodal Disease Measuring 15 mm or Greater | PET Positive Nodal Disease Measuring Less Than 15 mm | Patients Considered Resectable
Started | 15 | 0 (This arm was non-randomized and no enrolled patients fit the inclusion criteria for this group.) | 0 (This arm was non-randomized and no enrolled patients fit the inclusion criteria for this group.)
Completed | 13 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PET Positive Nodal Disease Measuring 15 mm or Greater | PET Positive Nodal Disease Measuring Less Than 15 mm | Patients Considered Resectable | Total
Number analyzed (Participants) | 13 | 0 | 0 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 7 |  |  | 7
  >=65 years | 6 |  |  | 6
Age, Continuous [Median (Full Range); unit: Years] | 62 [49 to 82] |  |  | 62 [49 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  |  | 4
  Male | 9 |  |  | 9
Region of Enrollment [Number; unit: participants]
  United States | 13 |  |  | 13

OUTCOME MEASURES:

1. Primary Outcome: Grade 3 or Higher Rate of Non-hematologic, Acute Treatment-related Toxicities
Time Frame: Six months after end of radiation therapy
Measure: Number; unit: participants
Arm/Group | PET Positive Nodal Disease Measuring 15 mm or Greater | PET Positive Nodal Disease Measuring Less Than 15 mm | Patients Considered Resectable
Number analyzed (Participants) | 13 | 0 | 0
participants | 1 |  |

2. Secondary Outcome: Percentage of Patients With Disease Control
Description: Disease control rate is defined as Complete Response (CR) + Partial Response (PR) + Stable Disease (SD). As per RECIST version 1.1, Complete Response (CR): Disappearance of all target lesions, Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study."), as accurate.
Time Frame: Following treatment every 6 months for 2 years, then annually for 4 years.
Population: Thirteen enrolled patients that completed treatment
Measure: Number; unit: percentage of participants
Arm/Group | PET Positive Nodal Disease Measuring 15 mm or Greater | PET Positive Nodal Disease Measuring Less Than 15 mm | Patients Considered Resectable
Number analyzed (Participants) | 13 | 0 | 0
percentage of participants | 69 |  |

3. Secondary Outcome: Percentage of Patients Alive at 5 Years
Time Frame: Five years following radiation treatment
Population: Thirteen enrolled patients that completed treatment.
Measure: Number; unit: percentage of patients
Arm/Group | PET Positive Nodal Disease Measuring 15 mm or Greater | PET Positive Nodal Disease Measuring Less Than 15 mm | Patients Considered Resectable
Number analyzed (Participants) | 13 | 0 | 0
percentage of patients | 69 |  |

4. Secondary Outcome: Feasibility, Safety and Efficacy of Delivering Proton Radiotherapy With Concomitant Chemotherapy
Time Frame: Weekly during treatment, then every 3 months for 1 year, every 4 months for 2 years, every 6 months for 2 years, then annually
Population: This data was not collected as study was terminated early.
Arm/Group | PET Positive Nodal Disease Measuring 15 mm or Greater | PET Positive Nodal Disease Measuring Less Than 15 mm | Patients Considered Resectable
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Correlation of Functional CT-PET Imaging With Treatment Outcomes
Time Frame: Prestudy, before surgery (if applicable) between days 18-22 if needed, then during follow-up every 6 months for 2 years, then annually for 4 years
Population: This data was not collected as study was terminated early.
Arm/Group | PET Positive Nodal Disease Measuring 15 mm or Greater | PET Positive Nodal Disease Measuring Less Than 15 mm | Patients Considered Resectable
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Cumulative adverse events assessed across all available post-treatment follow-up for each patient.
Arm/Group | PET Positive Nodal Disease Measuring 15 mm or Greater | PET Positive Nodal Disease Measuring Less Than 15 mm | Patients Considered Resectable
Serious Adverse Events (participants affected / at risk) | 2/13 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 13/13 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PET Positive Nodal Disease Measuring 15 mm or Greater (N=13) | PET Positive Nodal Disease Measuring Less Than 15 mm (N=0) | Patients Considered Resectable (N=0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 3
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 3
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 3
Weight loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PET Positive Nodal Disease Measuring 15 mm or Greater (N=13) | PET Positive Nodal Disease Measuring Less Than 15 mm (N=0) | Patients Considered Resectable (N=0)
Pain (General disorders) | 7 (7) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Radiation dermatitis (General disorders) | 4 (4) | 0 (0) | 0 (0)
White blood cell count (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Weight loss (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Alopecia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet count (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes